CLINICAL TRIAL: NCT00003183
Title: A Phase I/II Trial Using Weekly Mitoxantrone Chemotherapy and G-CSF for the Treatment of Metastatic Hormone Refractory Prostate Cancer
Brief Title: Mitoxantrone and G-CSF in Treating Patients With Metastatic Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hope Cancer Institute, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066007; HCRN-006; NCI-V98-1377
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Filgrastim; Mitoxantrone

INTERVENTIONS:
Biological: filgrastim
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with G-CSF may make tumor cells more sensitive to the chemotherapy drug and may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of mitoxantrone plus G-CSF in treating patients with metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Study the effectiveness of mitoxantrone in patients with metastatic, hormone refractory prostate cancer. II. Assess the side effects of mitoxantrone in this patient population. III. Determine whether filgrastim (granulocyte colony-stimulating factor; G-CSF) treatment can overcome chronic bone marrow suppression and facilitate a dose intensive mitoxantrone chemotherapy regimen in this patient population.

OUTLINE: This is a dose escalation study. Patients receive a 30 minute intravenous infusion of mitoxantrone once a week on day 1. On days 2-6 of each week, patients receive subcutaneous filgrastim (granulocyte colony-stimulating factor; G-CSF). Treatment continues for patients who respond to therapy and exhibit no disease progression. Dose escalation proceeds until the maximum tolerated dose (MTD) of mitoxantrone with G-CSF support is determined. The MTD is defined as the dose preceding that at which 2 or more patients experience dose limiting toxicity. After the MTD is determined, an additional 20-40 patients are enrolled at this dose level to examine their response to this therapy.

PROJECTED ACCRUAL: Approximately 12-24 patients will be accrued for the phase I portion of this protocol. An additional 20-40 patients may be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed hormone refractory adenocarcinoma of the prostate Metastatic disease required

PATIENT CHARACTERISTICS: Age: Not specified Performance status: SWOG 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: Absolute granulocyte count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL SGOT less than 2 times normal Renal: Creatinine less than 1.5 mg/dL Cardiovascular: Must have adequate cardiac function (LVEF at least 40%) Other: No other malignancy except skin lesions that have been completely excised No prior hypersensitivity to E. coli derived products

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: See Disease Characteristics At least 1 month since LHRH agonist and/or flutamide Radiotherapy: No concurrent radiotherapy No prior extensive radiotherapy (such as whole pelvic irradiation) Surgery: Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 1997-03

CONTACTS AND LOCATIONS:
Overall Officials: Raj Sadasivan, MD, PhD, Study Chair — Hope Cancer Institute, Inc.
Locations (2):
- United States (2):
  - Bethany Medical Center, Kansas City, Kansas
  - Heartland Cancer Research and Treatment Center, Kansas City, Kansas